CLINICAL TRIAL: NCT05498571
Title: Risk Prediction Model of Cardiovascular Events in Patients With Schizophrenia
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Shanghai Mental Health Center (Other)
Responsible Party: Sponsor
Other Study IDs: 2020-YJ13
Record Dates: First submitted 2021-11-21; First posted 2022-08-12 (Actual); Last update posted 2022-08-12 (Actual); Status verified 2022-04

CONDITIONS: Schizophrenia
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Schizophrenia Patients: We collect relevant information, review cardiovascular events in schizophrenia patients.

SUMMARY:
Schizophrenia is a serious mental illness that has a great impact on social function. Studies have evidenced that schizophrenia patients live 10-20 years less than general population.It mainly dues to high cardiovascular risk. How to improve patients' survival rates? At present, there is an objective model to assess cardiovascular risk among schizoprenia patients in England - PRIMROSE.But there is a lack of model for schizophrenia patients in china. In order to better guide clinical practice, we are now exploring a domestic cardiovascular risk prediction model to raise people's awareness.

DETAILED DESCRIPTION:
Schizophrenia is a common severe mental disorder with high rate of disability, which seriously affects patients' life.It is necessary to take long-term therapy to control symptoms or prevent recurrence. Studies have found that schizophrenia patients live on average ten to twenty-five years less than others. The main reason for high rates of mortality and disability is the high risk of cardiovascular events.There are few domestic large-scale studys on the risk of cardiovascular events in schizophrenia, thus they have not formed objective tools to assess cardiovascular risk. If this risk can be objectively assessed and predicted at an early stage, it is expected to reduce the risk of cardiovascular events and thus reduce mortality.At present, there are mature tools for assessing the risk of cardiovascular events in patients, such as Framingham, PRIMROSE, etc.The latter is the new tool for assessing cardiovascular events in patients with severe mental disorders. This study used a retrospective cohort design to collect the history of hospitalized schizophrenia patients within 2 years, collect relevant informations about cardiovascular events. The investigators validate the PRIMROSE model in China and explore the risk prediction model of cardiovascular events in schizophrenia patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients hospitalized before July 1, 2020；and hospitalized between July 1 2020-June 30, 2022；
* Meeting the ICD-10 diagnostic criteria for "Schizophrenia, Schizotypy, delusional disorder"or ICD-11 diagnostic criteria for "Schizophrenia and other Primary Mental Disorders";
* At least 2 doctors in charge of ward make definitive diagnoses;
* Age ≥18 years old, male and female are not limited.

Exclusion Criteria:

* Researchers consider patients unsuitable for the study;
* past history of cardiovascular disease (fatal and nonfatal cardiovascular events defined as myocardial infarction, Angina, coronary heart disease, coronary artery surgery, cerebrovascular accident and transient ischemic attack, peripheral arterial disease or revascularization) prior to antipsychotic therapy ;
* use of lipid lowering drugs or antiplatelet drugs, such as aspirin、statins ，prior to antipsychotic therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients hospitalized before July 1, 2020；and hospitalized between July 1 2020-June 30, 2022.The patients' diagnoses meet ICD-10 diagnostic criteria for "schizophrenia, schizophrenia, delusional disorder" or ICD-11 for "schizophrenia and other primary mental disorders".
Sampling Method: Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2021-12-01 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
cardiovascular events | 2-10 years
  Cardiovascular events end points were defined as the first occurrence of fatal or non-fatal cardiovascular events.They were collected and individually validated using data from the clinical diagnosis items, including data from emergency room visits, cardiology consultations, and tests (MRI,CT,ECG,Troponin I,Troponin T,coronary angiography etc). Fatal and non-fatal cardiovascular events are defined as myocardial infarction, Angina, coronary heart disease, coronary artery surgery, cerebrovascular accident and transient ischemic attack, peripheral artery disease or revascularization;cardiovascular and all-cause mortality.We need to record the time of the first cardiovascular events and diagnosis items.

CONTACTS AND LOCATIONS:
Overall Officials: Shengke Pan, Master, Study Director — Shanghai Mental Health Center
Locations (1):
- Shanghai Mental Health Center, Shanghai, Shanghai Municipality, China